CLINICAL TRIAL: NCT04793724
Title: Evaluation of Short-term Effect of Respiratory Physiotherapy Performed by Simeox on Lung Function in Patients With Primary Ciliary Dyskinesia - Randomised Cross-over Interventional Study
Brief Title: Respiratory Physiotherapy Performed by Simeox In Patients With Primary Ciliary Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Anna Chmelarova, Mgr, Principal Investigator, University Hospital, Motol
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PCD-375.2/20
Record Dates: First submitted 2021-02-22; First posted 2021-03-11 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: primary ciliary dyskinesia; respiratory physiotherapy; airway clearance techniques; lung function testing; ventilation inhomogeneity; nitrogen multiple breath washout test; spirometry; electric impedance tomography
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Intervention Model Description: First session - initial medical and physiotherapy assessment
  Second session - medical and physiotherapy assessment, respiratory physiotherapy with Simeox/PARI O PEP (according the randomization)
  Third session - medical and physiotherapy assessment, respiratory physiotherapy with Simeox/PARI O PEP (according the randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simeox first (Experimental): Patients who will undergo Simeox intervention first. After three months cross-over to PARI O PEP intervention.
  Interventions: Device: Simeox
- PARI O PEP first (Active Comparator): Patients who will undergo PARI O PEP intervention first. After three months cross-over to Simeox intervention.
  Interventions: Device: PARI O PEP

INTERVENTIONS:
Device: Simeox — A respiratory physiotherapy session with the Simeox device will be performed in accordance with the official PhysioAssist recommendations, which are;
  * clearance of the upper airways before the physiotherapy session
  * correct position of the mouthpiece in patient's mouth, with the lips placed on the thinnest part of the mouthpiece and the tongue positioned underneath the mouthpiece
  * slow nasal inhalation without too much recruitment of the inspiratory residual volume (IRV) and an exhalation with real deflation of the thorax
  * step-by-step shifting of the patient's tidal volume towards the expiratory residual volume (ERV), in order to target the most distal regions of the lungs
  * comfortable, relaxed sitting position with straightened spine
  * controlled cough, which will be encouraged only when it is productive
  Arms: Simeox first
Device: PARI O PEP — ACT with PARI O-PEP will be performed in an upright sitting position, using four positions of the device for the most effective clearance of mucus from the lungs. These positions will be:
  * horizontal;
  * low;
  * transition of the device from the low position to the horizontal position;
  * upside down.
  The mouthpiece will be placed between the patient's teeth as per standard procedure, and enclosed properly within the lips. Patients will perform slow and deep inhalation via the nose, then hold their breath for about 1 to 2 seconds at the end of inhalation. Exhalation will be performed slowly and completely into the PARI O-PEP through the patient's mouth. At the end of the session, the patient will perform "huffing" with the PARI O-PEP device in the upside down position in order to maintain open airways, and, if possible, expectoration sputum.
  Arms: PARI O PEP first

SUMMARY:
Primary ciliary dyskinesia (PCD) is characterized by impaired airway clearance and mucus stagnation. This results in recurrent upper and lower respiratory tract infections often leading to chronic inflammation and, if not treated early and properly, to irreversible functional and structural changes of the respiratory tract. As there is no causal treatment of PCD yet, airway clearance techniques (ACT) provide fundamental care for these patients.

Simeox is a new airway clearance device, recently developed by the French company PhysioAssist. This technology is based on pneumatic vibrations generated by the device itself. Vibrations are induced by rapidly alternating between atmospheric and negative pressure as the patient exhales, providing the most effective clearance of mucus from the lungs. Vibrations of different intensity and frequency are known to alter the rheological properties of mucus in the airways, whilst the negative pressure during exhalation helps to mobilise and drain the mucus to the central bronchi.

Although there have not yet been any evidence based papers published clarifying the effect of Simeox specifically in patients with PCD, using up-to-date information, experience, and positive feedback from our patients, we assume that there could be a significant benefit for the effectiveness of ACT.

DETAILED DESCRIPTION:
In this study the effectiveness of ACT will be evaluated based on the short-term effect(s) of respiratory physiotherapy with Simeox on changes in lung function and thoracic expansibility paediatric patients with PCD.

An interventional randomised non-inferiority crossover trial will be conducted in Motol University Hospital; the project was developed by the multidisciplinary team (MDT) of the Division of Paediatric Pulmonology of the Department of Paediatrics, 2nd Faculty of Medicine, Charles University in Prague and Motol University Hospital; and the Department of Rehabilitation and Sports Medicine, 2nd Faculty of Medicine, Charles University in Prague and Motol University Hospital.

Eligible patients will be randomly assigned into 2 arms - "Simeox-first group" and "Pari-O-PEP first" group. Randomisation will be done using computer generated code for each patient. The protocol will include 3 study visits - K0, K1 and K2 planned 3 months apart. After 6 months (second visit - K1), each patient will be switched to the other interventional group (crossed over). The first session (K0) includes an initial lung function assessment using spirometry, nitrogen-Multiple Breath Washout test (N2-MBW), Electrical Impedance Tomography (EIT), 6 Minute Walk Test (6 MWT), respiratory amplitudes (RA), and a theoretical introduction to therapy with the Simeox device. The second (K1) and third (K2) sessions will be interventional, including a respiratory physiotherapy session in between each measurement, excluding 6 MWT, which will be measured just once per session.

According to randomisation criteria, participants will initially undergo either physiotherapist-administered 20-minute ACT session using the Simeox device or 30-minute therapy with PARI O-PEP. In accordance with the rules for crossover study design, each patient will undergo therapy with both ACT devices, ideally within six-month duration of the study. These interventions will take place in between each measurement (spirometry, MBW, EIT, RA) during the second (K1) and the third (K2) session.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PCD confirmed by Transmission Electron Microscopy (TEM) analysis of ciliary ultrastructure showing clear structural axonemal defect and/or positive genetic testing for one (autosomal dominant) or two (autosomal recesive) PCD-causing mutations;
* age range 4 - 18 years;
* established chest physiotherapy with PARI O PEP

Exclusion Criteria:

* inability to undergo the assessment and intervention
* noncompliance and/or nonadherence

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Lung Clearance Index | Through study completion, an average of 1 year
  Ventilation Inhomogenity Assesment

SECONDARY OUTCOMES:
Change in Forced Residual Capacity (FRC) | Through study completion, an average of 1 year
  Volume of air present in the lungs at the end of passive expiration, in Litres [L].
Change in Forced Vital Capacity (FVC) | Through study completion, an average of 1 year
  Volume of air that can forcibly be blown out after full inspiration, in Litres [L]
Change in Forced Expiratory Volume in 1 second (FEV1) | Through study completion, an average of 1 year
  Volume of air exhaled in the first second during forced exhalation after full inspiration, in Litres per second [L/s]
Change in Maximal Expiratory Flow (MEF25-75) | Through study completion, an average of 1 year
  Volume of air where the certain amount (25-75%) of Forced Vital Capacity (FVC) remains to be exhaled, in Litres [L]
Change in Acinar airway inhomogeneity (Sacin) | Through study completion, an average of 1 year
  MBW indices reflecting ventilation inhomogeneity in the acinar airway region, in Litres [L]
Change in Conductive airway inhomogeneity (Scond) | Through study completion, an average of 1 year
  MBW indices reflecting ventilation inhomogeneity in the conductive airway region, in Litres [L]

OTHER OUTCOMES:
Change in Global Inhomogeneity (GI) Index | Through study completion, an average of 1 year
  Electrical Impedance Tomography parameter evaluating real-time spatial distribution of ventilation
Change in chest expansion measurement | Through study completion, an average of 1 year
  Chest expanson at axillary, mesosternal (mammary) and xiphosternal levels

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chmelarova, MD, Principal Investigator — Department of Rehabilitation and Sports Medicine, 2nd Faculty of Medicine
Locations (1):
- Motol University Hospital, Prague, Praha 5, Czechia

IPD SHARING:
Plan to Share IPD: No